CLINICAL TRIAL: NCT04736290
Title: The Effect of NLR and PLR on Perioperative Neurocognitive Disorders in Patients Undergoing Elective Non-cardiac Surgery Under General Anesthesia.
Brief Title: NLR and PRL in Neurocognitive Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Collaborators: University Hospital, Ioannina (Other); Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: NLR, PLR and NCD
Record Dates: First submitted 2020-10-24; First posted 2021-02-03 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Neurocognitive Disorders; Neutrophil-Lymphocyte Ratio; Platelet-Lymphocyte Ratio
Keywords: Neurocognitive disorders; Neutrophil-Lymphocyte ratio; Platelet-Lymphocyte ratio
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Noncardiac surgery: Calculation of the NLR and PLR in patients undergoing noncardiac surgery under general anesthesia
  Interventions: Other: NLR; Other: PLR

INTERVENTIONS:
Other: NLR — Calculation of NLR
Other: PLR — Calculation of PLR

SUMMARY:
Preliminary evidence suggest a possible relationship between Neutrophil-Lymphocyte Ratio (NLR) and Platelet-Lymphocyte Ratio (PLR) and perioperative neurocognitive disorders (NCD). We are going to investigate whether the values of NLR and PLR in patients undergoing elective non-cardiac surgery under general anesthesia, are related with increased risk of perioperative NCD.

DETAILED DESCRIPTION:
It is estimated that approximately 10% of elderly undergoing surgery will develop cognitive changes perioperatively, while in some reports the incidence rises up to 80%. Despite the reported high prevalence of perioperative neurocognitive disorders (NCD), their exact etiology is still largely unknown.

Preliminary evidence suggest a possible relationship between Neutrophil-Lymphocyte Ratio (NLR) and Platelet-Lymphocyte Ratio (PLR) and perioperative neurocognitive disorders (NCD). We are going to investigate whether the values of NLR and PLR in patients undergoing elective non-cardiac surgery under general anesthesia, are related with increased risk of perioperative NCD.

ELIGIBILITY:
Inclusion Criteria:

* 45 - 80 years
* American Society of Anesthesiologists physical status I to III
* elective general, urological, gynecological and orthopedic surgery under general anesthesia
* native speakers of the Greek language

Exclusion Criteria:

* refused to participate or sign the informed consent form
* had undergone surgery or anesthesia within the last 30 days
* had any prior or current history involving an affliction of the central nervous system
* were diagnosed with severe cognitive decline based on the 16 - item Informant Questionnaire on Cognitive Decline (IQCODE - 16)
* suffered from severe hearing or visual impairment
* any psychiatric disorder
* had a score >5 in the Geriatric Depression Scale (GDS - 15)
* or a score in females < 4 males < 2 in the Lawton - Brody Instrumental Activities of Daily Living Scale (I.A.D.L.)
* reported alcohol consumption > 35 units/week
* drug dependence
* had undergone previous neuropsychological testing
* Diabetes Mellitus type II with > 10 years of diagnosis
* Diabetes Mellitus type I
* Hemoglobin A1c (HbA1c) > 7.5%
* suffered from hemodynamical instability (> 20% alterations of blood pressure perioperatively)
* or desaturation (one or more events of SpO2 < 80% for more than 2 minutes) peri-operatively
* or blood loss of more than one unit

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 45 - 80 years old, ASA I-III undergoing elective general, urological, gynecological and orthopedic surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative neurocognitive disorders assessed with CAM | 1st postoperative day
  Incidence of POD assessed with CAM
Incidence of Postoperative neurocognitive disorders assessed with IQCODE-16 | 10th postoperative day
  Incidence of POCD assessed with IQCODE-16
Incidence of Postoperative neurocognitive disorders assessed with IQCODE-16 | 3 months postoperatively
  Incidence of POCD assessed with IQCODE-16
Incidence of Postoperative neurocognitive disorders assessed with IQCODE-16 | 6 months postoperatively
  Incidence of POCD assessed with IQCODE-16
Incidence of Postoperative neurocognitive disorders assessed with IQCODE-16 | 9 months postoperatively
  Incidence of POCD assessed with IQCODE-16

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, MD, PhD, Study Chair — Professor of Anesthesiology; Maria Ntalouka, MD, PhD, Principal Investigator — Consultant of Anesthesiology
Locations (1):
- University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: Undecided